CLINICAL TRIAL: NCT01747616
Title: Assessment of Safety and Tolerability of Chitosan-N-acetylcysteine Eye Drops in Subjects While Wearing Contact Lenses and Before Insertion of Contact Lenses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Croma-Pharma GmbH (Industry)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPHT-290311
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Dry Eye Syndrome
Keywords: Chitosan-N-Acetylcysteine; contact lenses; safety and tolerability
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 12 subjects wearing soft contact lenses (Experimental): The medical test device will be administered with the contact lenses inserted
  Interventions: Device: Chitosan-N-acetylcysteine eye drops (concentration of 0.1%); Other: Physiological saline solution
- 12 subjects wearing rigid contact lenses (Experimental): The medical test device will be administered with the contact lenses inserted
  Interventions: Device: Chitosan-N-acetylcysteine eye drops (concentration of 0.1%); Other: Physiological saline solution
- 12 subjects with soft contact lenses (Experimental): The medical test device will be administered before insertion of the contact lenses
  Interventions: Device: Chitosan-N-acetylcysteine eye drops (concentration of 0.1%); Other: Physiological saline solution
- 12 subjects with rigid contact lenses (Experimental): The medical test device will be administered before insertion of the contact lenses
  Interventions: Device: Chitosan-N-acetylcysteine eye drops (concentration of 0.1%); Other: Physiological saline solution

INTERVENTIONS:
Device: Chitosan-N-acetylcysteine eye drops (concentration of 0.1%) — 1 drop of the medical device in 1 randomly chosen eye
Other: Physiological saline solution — 1 drop as placebo in the other eye not receiving the medical device

SUMMARY:
The "dry eye syndrome" DES is a highly prevalent ocular disease, in particular in the elderly population. One mainstay of therapy for patients suffering from DES is the use of topically administered lubricants. However, despite many efforts, no "ideal" formulation has yet been found.

Recently, Croma Pharma has introduced chitosan-N-acetylcysteine eye drops, designed for treatment of symptoms related to DES. Chemically, chitosan is a polycationic biopolymer with favourable biological properties such as high biocompatibility and low toxicity. Additionally, the new formulation comprises N-acetylcysteine, which has been used in ophthalmology because of its mucolytic properties for several years. Based on theoretical considerations, one can hypothesize that the new chitosan derivative may show an increased adhesion to mucins of the ocular surface and may therefore be particularly beneficial in reducing the symptoms associated with DES. We have recently shown in a phase I trial that single instillation of chitosan-N-acetylcysteine eye drops is well tolerated in young healthy subjects.

However, no data is yet available about safety and tolerability of chitosan-N-acetylcysteine in subjects wearing contact lenses. This is of special interest because the tear film is critical to successful contact lens wear. Disturbances of the quantity or quality of the tear film results in intolerance of contact lens wear and possible damage to the ocular surface. This trial seeks to investigate the local tolerability and possible ocular discomfort of chitosan-N-acetylcysteine eye drops after repeated instillation .

ELIGIBILITY:
Inclusion Criteria:

* Regular contact lens wear since 3 years minimum
* Daily wearing time of the contact lens of 8 hours or more
* Good tolerability of the contact lenses without ocular discomfort or local signs of chemosis, conjunctival redness or other signs of intolerability as judged by the investigator.
* Subject willing to continue contact lens use for the study period
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings except ametropia

Exclusion Criteria:

* Participation in a clinical trial in the 3 weeks preceding the study
* Use of colored contact lenses
* Abuse of alcoholic beverages or other drugs
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-07; Primary Completion 2011-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Descriptive evaluation of ocular discomfort as assessed by the subjects | on 5 consecutive days before and after instillation of the eye drops

SECONDARY OUTCOMES:
Number of subjects with significant increase of redness | on 5 consecutive study days
Number of subjects experiencing adverse reactions | on 5 consecutive study days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Vienna, Austria